CLINICAL TRIAL: NCT01171131
Title: A Pilot Study to Identify Biomarkers Associated With Chronic TBI
Brief Title: A Pilot Study to Identify Biomarkers Associated With Chronic Traumatic Brain Injury
Acronym: Chronic TBI
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Georgene Hergenroeder, Associate Professor, Neurosurgery, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-09-0334
Record Dates: First submitted 2010-07-21; First posted 2010-07-28 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Saliva sample Blood sample (plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic TBI Patients - Non-penetrating: Chronic TBI patients should have a history of head trauma manifesting in one or more of the following:
  1. Loss of consciousness
  2. Post-traumatic amnesia
  3. Focal neurologic deficits, seizure
  4. Persistent symptoms of increased arousal (e.g. difficulty falling or staying asleep, anger and hypervigilance)
  5. Impairment in social, occupational, or other important areas of functioning (e.g. problems with work and relationships.) Patients will be excluded from the study if we are unable to obtain informed consent and if they are non-communicative (i.e. in a vegetative state).
  Interventions: Other: Blood/saliva sampling
- Chronic TBI Patients - Blast: Chronic TBI Blast injury patients should have a history of head trauma manifesting in one or more of the following:
  1. Loss of consciousness
  2. Post-traumatic amnesia
  3. Focal neurologic deficits, seizure
  4. Persistent symptoms of increased arousal (e.g. difficulty falling or staying asleep, anger and hypervigilance)
  5. Impairment in social, occupational, or other important areas of functioning (e.g. problems with work and relationships.) Patients will be excluded from the study if we are unable to obtain informed consent and if they are non-communicative (i.e. in a vegetative state).
  Interventions: Other: Blood/saliva sampling
- Healthy Volunteers: Healthy volunteers include gender, age and race matched volunteers able to provide informed consent who have,
  1. No significant medical history
  2. Take no medications (other than birth control pills)
  3. Fever free
  4. No history of head trauma or recent injury/infection
  5. No history of neurological or psychiatric disorders or alcohol or drug dependency.
  Interventions: Other: Blood/saliva sampling

INTERVENTIONS:
Other: Blood/saliva sampling — one-time blood sample (~ 1 TBS) and saliva sample (~ 1 tsp)

SUMMARY:
The aim of this research is to determine if the biological fluids (blood/saliva) from chronic brain-injured patients (both blast and non-penetrating TBI) contain reproducible protein markers. To accomplish this two populations of chronic TBI patients who are receiving treatment at The Institute for Research and Rehabilitation (TIRR): blast injury victims and non-penetrating TBI will be studied. Using multiple proteomic approaches including mass spectrometry, multiplex ELISAs, and antibody microarrays, as well as RNA profiling, the investigators aim to identify biomarkers in the blood/saliva of patients suffering from chronic TBI and to determine the similarities/differences between the blast and non-penetrating injury groups. Identification of these biochemical changes will give insight into the long-lasting changes associated with head injury, and may identify new targets for treating the associated pathologies.

ELIGIBILITY:
Chronic TBI patients:

Inclusion Criteria

Have a history of head trauma manifesting in one or more of the following:

* Loss of consciousness
* Post-traumatic amnesia
* Focal neurologic deficits, seizure
* Persistent symptoms of increased arousal (e.g. difficulty falling or staying asleep, anger and hypervigilance)
* Impairment in social, occupational, or other important areas of functioning (e.g. problems with work and relationships.)

Exclusion Criteria

Inability to obtain informed consent and if they are non-communicative (i.e. in a vegetative state).

Healthy volunteers:

Inclusion Criteria

* No significant medical history
* Take no medications (other than birth control pills)
* Fever free
* No history of head trauma or recent injury/infection
* No history of neurological or psychiatric disorders or alcohol or drug dependency.

Exclusion Criteria

* Inability to provide informed consent
* age/gender match not available in TBI cohort

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TIRR Clinics
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2016-03-03 (Actual)

PRIMARY OUTCOMES:
Proteomic analysis of plasma | average of 6 months post injury
  The aim is to identify biomarkers in the blood of patients suffering from chronic TBI and to determine the similarities/differences between the blast and non-penetrating injury groups.

SECONDARY OUTCOMES:
Proteomic analysis of saliva | average of 6 months post injury
  The aim is to identify biomarkers in the saliva of patients suffering from chronic TBI and to determine the similarities/differences between the blast and non-penetrating injury groups.

CONTACTS AND LOCATIONS:
Overall Officials: Georgene Hergenroeder, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- TIRR, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data